CLINICAL TRIAL: NCT01160796
Title: Study of the Efficacy and Safety of Treatment With Total Freeze-dried Culture of Lactobacillus Casei Var. Rhamnosus (Lcr35®) Administered Intravaginally in the Prevention of Bacterial Vaginosis. Randomized, Phase III, Multi-centre, Double-blind, Placebo-controlled Superiority Trial
Brief Title: Lcr35® for Bacterial Vaginosis Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Lyocentre (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PREVA
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lcr35® (Experimental)
  Interventions: Drug: Lcr35®
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — 1x14-day course of treatment during 4 cycles
  Arms: placebo
Drug: Lcr35® — 1x14-day course of treatment during 4 cycles
  Arms: Lcr35®

SUMMARY:
This is a national, multi-centre, randomized, double-blind placebo-controlled, phase III superiority trial.

The main objective of the trial is to assess the efficacy of Lcr35® by comparing the mean time before the onset of the first clinical recurrence confirmed by laboratory tests in patients with bacterial vaginosis treated with Lcr35® versus placebo.

Patients with bacterial vaginosis will be enroll by private gynecologists. Each patient will receive a treatment for the initial episode(Metronidazole)and a treatment to prevent the recurrence of bacterial vaginosis (Lcr35®).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with a symptomatic vaginosis characterised by the presence of the following 3 clinical criteria (among the 4 Amsel criteria) at V1:

  * greyish uniform vaginal discharge,
  * characteristic "rotten fish" smell caused by the spontaneous release of amine or during the potassium test or "sniff test",
  * vaginal pH greater than 4.5.
* Patient with a Nugent score ≥ 7 (using the sample taken at V1).
* Patient clinically cured (none of the 3 Amsel criteria) after a 7-day course of Metronidazole (Flagyl®) Female.
* Patient over 18 years of age.
* For women with childbearing potential:

  * negative urine pregnancy test,
  * use of a contraceptive method deemed effective by the Investigator (excluding spermicides).
* Patient having received information and voluntarily signed a written Informed Consent Form.
* Patient covered by a national insurance scheme.

Exclusion Criteria:

* Presence of a yeast infection that is bacterial (other than vaginosis) or viral in origin presumed or proven to be gynaecologically-linked, whether or not treated within the month preceding inclusion or present at the time of inclusion.
* Presence of an existing gynaecological infection that may interfere with the assessment of the trial treatment(fibroma, severe dysplasia of the cervix or in situ carcinoma, invasive carcinoma, intra-epithelial cervical neoplasia, squamous intra-epithelial lesions etc.)
* Antibiotics or antifungals taken by general route during the month preceding the screening visit, excluding treatment for an earlier episode of vaginosis.
* Use of probiotics in the month preceding the screening visit, excluding treatment for an earlier episode of vaginosis.
* Use of intravaginal antiseptics in the month preceding the screening visit, excluding treatment for an earlier episode of vaginosis.
* Use of prebiotics (acidifiers) during the two weeks preceding the screening visit.
* Use of products containing topical oestrogens during the month preceding the screening visit.
* Allergy to one of the active ingredients or one of the excipients in the products.
* patient in post-menopausal time
* Patient unable to comply with the constraints of the Protocol.
* Breastfeeding patient.
* Patient with menstrual bleeds lasting more than 12 days a month.
* Patient having taken part in a clinical trial in the 3 months preceding inclusion in the present Protocol.
* Patient with a severe acute or chronic disease deemed by the Investigator to be incompatible with participation in the trial, or a serious infection that is life-threatening in the short term.
* Immuno-suppressed patient.
* Patient presenting with a previous illness which, according to the Investigator, is likely to interfere with the results of the trial or expose the patient to an additional risk.
* Patient linguistically or mentally unable to understand and sign the Informed Consent Form.
* Patient deprived of her liberty by order of the Courts or civil authorities or subject to a guardianship order.
* Patient likely not to comply with treatment.
* Patient unable to be contacted in the case of an emergency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
mean time before the onset of first clinical recurrence confirmed by laboratory tests | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Lyocentre, Aurillac, France